CLINICAL TRIAL: NCT04721665
Title: German SLD-Registry Characterization of Patients with Steatotic Liver Disease (SLD) in Germany - Phase 1 (observation of the Natural Course)
Brief Title: German SLD-Registry (Deutsches SLD-Register)
Status: Recruiting | Type: Observational
Sponsor: Leberstiftungs-GmbH Deutschland (Industry)
Responsible Party: Sponsor
Other Study IDs: NAFLD_01
Record Dates: First submitted 2020-11-30; First posted 2021-01-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Steatotic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SLD patients: No intervention

SUMMARY:
Characterization of patients with steatotic liver disease (SLD)

The German SLD-Registry (Deutsches SLD-Register) a project of the German Liver Foundation (Deutsche Leberstiftung), managed by Leberstiftungs-GmbH Deutschland.

The German NAFLD-Registry is financially supported by: Advanz Pharma Specialty Medicine Deutschland GmbH und Gilead Sciences GmbH (Grant to German Livber Foundation) sowie Novo Nordisk Pharma GmbH (directly via Leberstiftungs-GmbH).

DETAILED DESCRIPTION:
The following data can be documented:

* physical examination and vital parameters (e.g. age, weight)
* comorbidities (e.g. diabetes mellitus, cardiovascular disease)
* comedication (treatment of comorbidities related to SLD)
* laboratory values (e.g. liver function tests, creatinine)
* genetic variants (e.g. PNPLA3)
* liver diagnostics (e.g. histological findings, sonographic findings)
* lifestyle (alcohol consumption, physical activity)
* health related quality of life (SF-36 questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* diagnosed SLD based on the following criteria:

  1. typical finding of hepatic steatosis (abdominal ultrasound and/or pathological CAP value (latter is optional)
  2. Evaluation of SLD degree by NAFLD Fibrosis score and/or FIB-4-Index and/or transient elastography
  3. Evaluation of metabolic syndrome
* credible assessment of alcohol consumption
* written informed consent

Exclusion Criteria:

* patients with other hepatologic diseases (chronically viral, metabolic, autoimmune origin
* patients receiving hepatotoxic medications over a longer period (e.g. methotrexate, amiodarone, longterm NSAR intake)
* malignant disease with a life expectancy <12 months
* participation in clinical interventional/pivotal studies
* inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of patients to be enrolled with SLD is limited to 10,000.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2036-11-30 (Estimated); Study Completion 2036-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression of liver fibrosis | through study completion, an average of 1 year
  Fibrosis stage is measured by elastography (elastometry kPa value).
Activity of metabolic dysfunction-associated steatohepatitis (MASH) | through study completion, an average of 1 year
  Activity is measured via histology (NAFLD activity score represents the sum of scores for steatosis, lobular inflammation, and ballooning, and ranges from 0-8.)
Cardiovascular events | through study completion, an average of 1 year
  The onset of the clinical outcome cardiovascular events (yes/no)
Tumor diseases | through study completion, an average of 1 year
  The onset of the clinical outcome tumor diseases (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zeuzem, Prof. Dr., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (14):
- Germany (14):
  - Infektiologisches Zentrum Steglitz, Berlin
  - Leber- und Studienzentrum Checkpoint, Berlin
  - MVZ für Gastroenterologie am Bayerischen Platz, Berlin
  - Praxis für Innere Medizin mit Schwerpunkt Gastroenterologie Dr. med. Jeannette Schwenzer, Berlin
  - MVZ Viszeralmedizin GmbH, Cologne
  - Praxis Ludwig und Dikopoulos, Dornstadt
  - Fachinternistische Schwerpunktpraxis, Hamburg
  - Gastroenterologische Studiengesellschaft Herne, Herne
  - Leberstudienzentrum Kiel, Kiel
  - Eugastro GmbH, Leipzig
  - MVZ Dres. Eisenbach,Simon, Schwarz GbR, Leverkusen
  - Praxis Dr. med. Kerstin Stein, Magdeburg
  - CIM GmbH, Münster
  - St. Josefs-Hospital Medizinische Klinik II, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related information on the registry — https://www.deutsches-nafld-register.de/